CLINICAL TRIAL: NCT05432167
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group, Dose-Ranging Study to Evaluate CIN-107 for the Treatment of Patients With Uncontrolled Hypertension and Chronic Kidney Disease
Brief Title: A Study to Evaluate CIN-107 for the Treatment of Patients With Uncontrolled Hypertension and Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIN-107-123; D6972C00001 (Other: AstraZeneca)
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Uncontrolled Hypertension; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose CIN-107 (Experimental): Patients will take oral tablets of CIN-107 for 26 weeks. The dose strength may be titrated within 6 weeks.
  Interventions: Drug: CIN-107
- High dose CIN-107 (Experimental): Patients will take oral tablets of CIN-107 for 26 weeks. The dose strength may be titrated within 6 weeks.
  Interventions: Drug: CIN-107
- Placebo (Placebo Comparator): Patients will take oral tablets of Placebo for 26 weeks. The dose strength may be titrated within 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIN-107 — Patients will take CIN-107 tablets by mouth once daily.
  Arms: High dose CIN-107; Low dose CIN-107
Drug: Placebo — Patients will take placebo tablets by mouth once daily.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of CIN-107 for the treatment of hypertension in patients with uncontrolled hypertension (uHTN) and Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled will evaluate the efficacy and safety of CIN-107 in patients with uHTN and CKD. Approximately 200 patients will be randomized in a 1:1:1 ratio into 1 of the 3 treatment groups (placebo, low dose treatment strategy and high dose treatment strategy).

The study will consist of the following 3 periods:

* A Screening Period of up to 5 weeks;
* A Double-Blind Treatment Period of 26 weeks; and
* A Follow-Up Period of 2 weeks.

Patients will complete the study in approximately 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Has a mean seated SBP ≥ 140 mmHg.
* Has a prior diagnosis of mild-to-severe CKD.
* Has an elevated UACR.
* Is currently taking an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) at the maximum tolerated daily dose.

Exclusion Criteria:

* Have a documented diagnosis of type 1 diabetes.
* Are not willing or not able to discontinue a mineralocorticoid receptor antagonist (MRA) or a potassium sparing diuretic as part of an existing antihypertensive regimen.
* Have a single occurrence of mean seated SBP >180 mmHg or DBP >110 mmHg during the Screening Period.
* Has a body mass index (BMI) >50 kg/m^2.
* Has documented bilateral clinically relevant renal artery stenosis of ≥70%.
* Has had dialysis for acute kidney injury/acute renal failure within 12 weeks prior to the Screening Period or has a planned dialysis or kidney transplantation during the course of the study.
* Has known documented chronic heart failure New York Heart Association Class III or Class IV and/or hospitalization for heart failure within 6 months of Screening.
* Has had a stroke, transient ischemic attack, hypertensive encephalopathy, acute coronary syndrome, or hospitalization for heart failure within 6 months of Screening.
* Has known current severe left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy and/or severe aortic valvular disease.
* Has planned any major cardiac surgery during the study or had major cardiac surgery within 6 months of Screening.
* Has had a prior solid organ transplant or cell transplant.
* Has a known hypersensitivity to CIN-107 or drugs of the same class
* Has received immunotherapy for treatment of CKD within 6 months of Screening.
* Has any clinically relevant medical or surgical conditions including unstable conditions and/or conditions requiring regular transfusion or treatment with systemic immunosuppressants, including corticosteroids.
* Serum potassium <3.5 mEq/L or >5.0 mEq/L
* Serum sodium <135 mEq/L
* Serum aspartate aminotransferase or alanine aminotransferase >3 × upper limit of normal (ULN); or Total bilirubin >2 × ULN, unless due to Gilbert's syndrome.
* GFR is < 25 or > 75 mL/min/1.73 m2
* Has uncontrolled diabetes with glycosylated hemoglobin >10.5%.
* Is positive for Human immunodeficiency disease (HIV) antibody, hepatitis B surface antigen, or hepatitis C virus Ribonucleic acid (RNA).
* Has typical consumption of >14 alcoholic drinks weekly.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (68):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Beverly Hills, California
  - Research Site, Chula Vista, California
  - Research Site, Fountain Valley, California
  - Research Site, Granada Hills, California
  - Research Site, Lancaster, California
  - Research Site, Lincoln, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Northridge, California
  - Research Site, Panorama City, California
  - Research Site, Pomona, California
  - Research Site, Rancho Cucamonga, California
  - Research Site, Riverside, California
  - Research Site, San Dimas, California
  - Research Site, South Gate, California
  - Research Site, Tarzana, California
  - Research Site, Vacaville, California
  - Research Site, Victorville, California
  - Research Site, Arvada, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Hollywood, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Nampa, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Silver Spring, Maryland
  - Research Site, New Bedford, Massachusetts
  - Research Site, Flint, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Olive Branch, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Trenton, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Oxford, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Bethany, Oklahoma
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Paris, Texas
  - Research Site, Red Oak, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Alexandria, Virginia
  - Research Site, Burke, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Kingwood, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Dwyer JP, Maklad N, Vedin O, Monyak J, Myte R, Chertow GM, Heerspink HJL, Little DJ. Efficacy and Safety of Baxdrostat in Participants with CKD and Uncontrolled Hypertension: A Randomized, Double-Blind, Placebo-Controlled Trial. J Am Soc Nephrol. 2025 Sep 6. doi: 10.1681/ASN.0000000849. Online ahead of print. No abstract available. PMID 40913594
- [Derived] Townsend RR. Blocking Aldosterone Synthesis: Whose BrigHTN Idea Was That? Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1631-1633. doi: 10.2215/CJN.0000000000000265. Epub 2023 Jul 24. No abstract available. PMID 37490693
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-123&attachmentIdentifier=b12e7f74-0d50-4db5-a61a-d7c873db4754&fileName=CSP_CIN-107-123_PDFA_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-123&attachmentIdentifier=eac2398c-f0a8-4811-8d5f-ba17e99f4de4&fileName=SAP_CIN-107-123_PDFA_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-123&attachmentIdentifier=1b1f4d13-ac35-470f-8f10-70eb60638d80&fileName=CSR_Synopsis_CIN-107-123_PDFA_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 29 April 2022 to 02 May 2024 at 78 sites in the United States.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- CIN-107 Low Dosing Strategy Group: Participants received oral tablets of low dose strengths of CIN-107 for 26 weeks.
- CIN-107 High Dosing Strategy Group: Participants received oral tablets of high dose strengths of CIN-107 for 26 weeks.
- Placebo: Participants received oral tablets of Placebo for 26 weeks.
Period: Overall Study
Arm/Group | CIN-107 Low Dosing Strategy Group | CIN-107 High Dosing Strategy Group | Placebo
Started | 65 | 64 | 66
Completed | 53 | 54 | 51
Not Completed | 12 | 10 | 15
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Lost to Follow-up | 3 | 3 | 2
Not completed — Inclusion/exclusion criteria not met | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 11
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (ITT) included all participants randomized into the study. Treatment classification was based on the randomized treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CIN-107 Low Dosing Strategy Group | CIN-107 High Dosing Strategy Group | Placebo | Total
Number analyzed (Participants) | 65 | 64 | 66 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 67.2 (12.63) | 66.5 (11.02) | 65.6 (10.79) | 66.4 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 19 | 63
  Male | 42 | 43 | 47 | 132
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4 | 3 | 5 | 12
  Race: Black or African American | 19 | 24 | 20 | 63
  Race: White | 41 | 34 | 38 | 113
  Race: Other | 0 | 1 | 2 | 3
  Race: Not Reported | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated Systolic Blood Pressure (SBP) of Pooled CIN-107 and Placebo
Description: Mean change in seated SBP from baseline to Week 26 of pooled CIN-107 and placebo was assessed.
Time Frame: At Week 26
Population: Modified Intent-to-treat (mITT) population included all participants in the ITT population who received at least 1 dose of any study drug.
  Here, 'overall number of participants analyzed' means the number of participants with non-missing data.
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Groups:
- CIN-107 Treatment Groups Pooled: Participants received oral tablets of high and low doses of CIN-107 for 26 weeks.
Arm/Group | CIN-107 Treatment Groups Pooled | Placebo
Number analyzed (Participants) | 105 | 48
Millimeters of mercury (mmHg) | -15.22 (1.532) | -7.15 (2.231)
Statistical Analysis 1: Comparison: CIN-107 Treatment Groups Pooled vs Placebo; The analysis was performed using a mixed-effect model for repeated measures including fixed effects for treatment, visit, stratification variables (SGLT2 inhibitor use and CKD category), and the treatment-by-visit interaction, along with a covariate of the baseline seated SBP value and the baseline seated SBP by visit interaction; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -8.08, 95% CI 2-sided [-13.36 to -2.79], Standard Error of Mean 2.676

2. Secondary Outcome: Change From Baseline in SBP in CIN-107 Compared to Placebo in Participants Assigned to the High-dose Strategy Group
Description: Mean change in seated SBP from baseline to Week 26 of high-dose CIN-107 dosing group and placebo was assessed.
Time Frame: At Week 26
Population: mITT population included all participants in the ITT population who received at least 1 dose of any study drug.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | CIN-107 High Dosing Strategy Group | Placebo
Number analyzed (Participants) | 63 | 64
mmHg | -14.37 (2.117) | -7.16 (2.233)
Statistical Analysis 1: Comparison: CIN-107 High Dosing Strategy Group vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = -7.22, 95% CI 2-sided [-13.24 to -1.19], Standard Error of Mean 3.051

3. Secondary Outcome: Change From Baseline of SBP in CIN-107 Compared to Placebo in Participants Assigned to the Low-dose Strategy Group
Description: The mean change in seated SBP from baseline to Week 26 of low-dose CIN-107 dosing group and placebo was assessed.
Time Frame: At Week 26
Population: mITT population included all participants in the ITT population who received at least 1 dose of any study drug.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | CIN-107 Low Dosing Strategy Group | Placebo
Number analyzed (Participants) | 65 | 64
mmHg | -16.14 (2.186) | -7.16 (2.233)
Statistical Analysis 1: Comparison: CIN-107 Low Dosing Strategy Group vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -8.99, 95% CI 2-sided [-15.10 to -2.87], Standard Error of Mean 3.098

4. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: The safety and tolerability of CIN-107 in participants with uncontrolled hypertension (uHTN) and chronic kidney disease (CKD) was assessed.
  Adverse events of special interest (AESI) include any hypotension events, abnormal potassium or sodium laboratory values that require clinical intervention.
Time Frame: From randomization (Day 1) until the end of Follow up period (approximately 8 months)
Population: Safety population included all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CIN-107 Low Dosing Strategy Group | CIN-107 High Dosing Strategy Group | Placebo
Number analyzed (Participants) | 65 | 63 | 64
Participants
  All TEAEs | 48 | 52 | 35
  All TEAEs, related to treatment | 23 | 31 | 14
  Any TEAE with outcome = Death | 0 | 0 | 0
  Any TEAE with outcome = Death, related to treatment | 0 | 0 | 0
  Any TEAE leading to dose interruption | 20 | 23 | 13
  Any TEAE leading to dose interruption, related to treatment | 10 | 10 | 4
  Any TEAE leading to discontinuation of treatment | 10 | 11 | 5
  Any TEAE leading to discontinuation of treatment, related to treatment | 7 | 8 | 3
  Any TEAE leading to discontinuation of study | 0 | 2 | 1
  Any TEAE leading to discontinuation of study, related to treatment | 0 | 1 | 1
  All treatment emergent serious adverse events (TESAEs) | 7 | 5 | 2
  All TESAEs, related to treatment | 2 | 1 | 1
  Any TESAE with outcome = Death | 0 | 0 | 0
  Any TESAE with outcome = Death, related to treatment | 0 | 0 | 0
  Any TESAE leading to dose interruption | 2 | 1 | 1
  Any TESAE leading to dose interruption, related to treatment | 0 | 0 | 1
  Any TESAE leading to discontinuation of treatment | 2 | 2 | 1
  Any TESAE leading to discontinuation of treatment, related to treatment | 2 | 1 | 0
  Any TESAE leading to discontinuation of study | 0 | 1 | 0
  Any TESAE leading to discontinuation of study, related to treatment | 0 | 0 | 0
  Treatment emergent AESIs | 11 | 12 | 4

ADVERSE EVENTS:
Time Frame: From randomization (Day 1) until the end of Follow up period (approximately 8 months)
Description: Safety population included all participants who received at least one dose of any study drug.
Arm/Group | CIN-107 Low Dosing Strategy Group | CIN-107 High Dosing Strategy Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 7/65 | 5/63 | 2/64
Other Adverse Events (participants affected / at risk) | 47/65 | 52/63 | 35/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIN-107 Low Dosing Strategy Group (N=65) | CIN-107 High Dosing Strategy Group (N=63) | Placebo (N=64)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIN-107 Low Dosing Strategy Group (N=65) | CIN-107 High Dosing Strategy Group (N=63) | Placebo (N=64)
Hyperkalaemia (Metabolism and nutrition disorders) | 21 (30) | 32 (52) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 11 (14) | 15 (20) | 5 (7)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 4 (4) | 5 (6)
Lipase increased (Investigations) | 2 (3) | 3 (3) | 1 (1)
Blood potassium increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QRS complex shortened (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT interval abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (2) | 2 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Renal impairment (Renal and urinary disorders) | 2 (2) | 5 (5) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (3) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) | 2 (3)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Overflow diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca.

DOCUMENTS (2):
  • Study Protocol (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT05432167/Prot_002.pdf
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT05432167/SAP_003.pdf